CLINICAL TRIAL: NCT01983852
Title: Paediatric End of Life Care Needs in Switzerland
Acronym: PELICAN
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: University Children's Hospital, Zurich (Other); University Children's Hospital Bern (Unknown); University Children's Hospital Basel (Other); Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other); University of Lausanne (Other); Ospedale Regionale Bellinzona e Valli (Other)
Responsible Party: Principal Investigator, Eva Cignacco, PD, Phd, University of Basel
Other Study IDs: PELICAN_2012_2015; KFS-3008-08-2012 (Other Grant/Funding Number: KFS-3008-08-2012)
Record Dates: First submitted 2013-10-31; First posted 2013-11-14 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Paediatric Palliative Care
Keywords: End of Life Care; Paediatric; Experiences; Needs; Current Practices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children during End of Life Care

SUMMARY:
Background Children living with life-limiting conditions have always been part of the health care system. Although there have been dramatic improvements in medical care, hundreds of children continue to die annually. The field of paediatric palliative care (PPC) and end-of-life (EOL) care is based on the principle that an interdisciplinary team should care for patients and their families. However, evidence on how to provide optimal PPC and EOL care covering the needs of children and their families is scarce and lags substantially behind that in the adult world. Few is known on how EOL care - defined as the last four weeks of life in this study - is presently provided in the Swiss health setting. The presented study Paediatric End-of-LIfe CAre Needs in Switzerland [PELICAN]) covers paediatric EOL care and will contribute to a comprehensive understanding of EOL care in Switzerland by analysing retrospectively medical charts of children/young people between 0 - 18 years who died in the years 2010 and 2011 in Switzerland. A survey instrument will be developed and pilot tested to assess the perspectives of families who have experienced the loss of a child. After the development pilot testing and adaptation of the instrument a survey with parents who lost a child in the years 2010 and 2011 will take place. Furthermore, the experiences and needs of health professionals working in the field of pediatric EOL will be explored.

DETAILED DESCRIPTION:
Children living with life-limiting conditions have always been part of the health care system. Although there have been dramatic improvements in medical care, hundreds of children continue to die annually. In Switzerland, approximately 400 children (0 to 14 years of age) die each year, about three quarters of those due to a medical condition. Infant deaths account for approximately half of the deaths during childhood and are mostly due to perinatal conditions. Complex chronic conditions such as congenital and chromosomal abnormalities, diseases of the nervous system, cancer and cardiac conditions constitute the most important group of disease-related death in childhood. This underlines the rationale to include children who died due to an oncological, cardiological or neurological disease or during the neonatal period (from birth up to four weeks of life) in this study.

Characteristics of End-of-Life (EOL) Care and death during childhood When the burden of disease and poor quality of life outweigh the potential benefit of disease related treatments, the focus of care shifts towards preparing for an anticipated death and managing the end stage of a terminal medical condition. Through a process of literature review, clinician and parent surveys and interviews, six domains of high-quality, family-centred EOL care have been identified: 1) support of the family unit [the unit of care is the child and the family, whereas family is defined as those who provide comfort to the child, regardless of genetic relationship]; 2) communication with the child and the family about treatment goals and plans; 3) ethics and shared decision making; 4) relief of pain and other symptoms; 5) continuity of care; and 6) grief and bereavement support. Nonetheless, questions about how to best provide EOL care for dying children remain inadequately answered, as there are no systematic studies on EOL care in children. Apart from that, there is a lack of interventional studies, which are very difficult to perform in such an ethical sensitive field of care.

Dying at home is often associated with good quality of EOL care and a "good death" and the view that most patients prefer to die at home is commonly accepted. In reality, paediatric home death rates, although growing, have remained low at 20% between 1999-2003 in the United States. There is some evidence that parents whose child died at home from cancer show lower levels of grief-related symptoms and psychological distress. However a recent study by Dussel et al. showed that the opportunity to plan the place of death is associated with outcomes consistent with high-quality EOL care, and thus may represent a more relevant outcome than the actual place of death. Neonatal intensive care units (NICU) and paediatric intensive care units (PICU) play a particular important role in EOL care as they are a place where a high percentage of paediatric patients die. For newborns, only rarely exists a valuable alternative to the NICU. It is important to know when, where and under which circumstances children die, and to know the impact of characteristics of death on the overall satisfaction of parents with EOL care. No data about current practice of EOL care and the characteristics of the child's death exists for Switzerland.

Parents' perspectives on EOL care of their dying child EOL care of these vulnerable patients and families demands a comprehensive approach that includes the need for health care professionals to understand the illness experience from the perspective of the dying child and its family. Guidelines for EOL care of children are focused on effective symptom management and clear communication, yet parents' values for EOL care are still partly unknown. There is overwhelming evidence that communication is central to the concerns of parents and it is the principle determinant of high-quality care. Professional support in the last four weeks of life was a significant factor associated with having worked through their grief for parents who lost a child to cancer. Recently, a qualitative study was conducted in Switzerland exploring the perceptions and needs of families who cared for a child with life-limiting disease. Shortcomings were demonstrated and basic needs of affected families such as psychosocial support, coordination of care and bereavement support were outlined. To get a comprehensive picture of parental perspectives a population-based assessment is needed to quantify and explain their experiences and needs. This is only achievable through questionnaire survey and interviews with parents. As showcased by a systematic literature review, no tools exist to assess the needs of parents whose children died (i.e., in PICU). Questionnaires have been used in the field of EOL care, but none fits the unique requirements of the PELICAN research programme covering four distinct diagnostic groups.

Perspectives of health care professionals Several studies reported on barriers in the provision of paediatric palliative care (PPC) and EOL care. To develop a successful program for PPC and EOL care in Switzerland, barriers and gaps of knowledge, professional attitudes, skills and structural preconditions need to be perceived. In Germany, a recent study revealed significant shortcomings in financing of specialist nursing home care that necessarily includes funding of coordination and case-management. Another issue was the required openness towards PPC and EOL care from professionals, particularly physicians that is a prerequisite for family-centred EOL care. There are only few articles describing how to assess attitudinal, educational and institutional issues in professionals. One study from Australia developed a questionnaire to measure barriers and facilitators of palliative care in neonatal nursing. From 645 neonatal nurses 57% reported staffing as adequate to support a palliative care practice, 57% reported that the environment of their unit was not conducive to provide palliative care to dying infants, while 62% felt that they often went beyond of what they estimated comfortable when providing technological life support to dying new-borns. A study from the United States described barriers to EOL care for children and their families, as perceived by paediatric health care providers. An important finding was, that perceived barriers to paediatric EOL care differed from those impeding adult EOL care. Commonly perceived barriers to paediatric EOL care involved uncertainties in prognosis and discrepancies in treatment goals between staff members and family members. Improved staff education may help to overcome some of these obstacles; however, the most effective methods of improving nurses' and physicians' competences in PPC and EOL care remains to be established. In Switzerland, a recent study with 76 paediatric health care professionals explored expectations on specialised PPC teams. From the perspectives of non-specialised care providers the tasks would particularly encompass the coaching of attending teams, coordination of care, symptom control, and direct support of affected families during and beyond the illness of their child. More systematic data and specific knowledge of the situation in Switzerland is urgently needed to meet the needs of health care professionals and provide them with adequate knowledge on how to best provide EOL care.

Rationale The field of paediatric palliative care (PPC) and EOL care is based on the principle that an interdisciplinary team should care for patients and their families. However, evidence on how to provide optimal PPC and EOL care covering the needs of children and their families is scarce and lags substantially behind that in the adult world. Few is known on how EOL care - defined as the last four weeks of life in this study - is presently provided in the Swiss health setting. Generalizability of study results from other countries is limited. In contrast to many other countries, there are no paediatric hospices in Switzerland. EOL care is challenging for health professionals. Being aware of current practices and the parents' perspectives helps showing the difference that good quality EOL care and support can make to a family losing their child. To meet the parents' values for care, it is important to assess the needs of this vulnerable group directly. Diverse medical conditions imply different needs. This circumstance demands the development of a survey instrument that matches specific diagnoses and their specific illness. In addition to the parents', the evaluation of perspectives and needs of health professionals is important for the development of services which should be used by non-specialized care providers. The combination of a qualitative and quantitative approach enhances a comprehensive discovery of this existentially high subjective human experience.

Study Aims The overarching aim of the present study is to provide comprehensive information and understanding about the current practices of EOL care in the paediatric setting in Switzerland (hospital and community health care), about parental perspectives and the perspectives of the health care professionals in order to formulate required steps to improve care during this highly vulnerable and critical phase of life.

Specific aims are stated as follows:

PELICAN I - Aims.

1. Description of current practice of EOL care in Switzerland for children/adolescents who died from a cardiological, neurological or oncological disease, or who died during the neonatal period
2. Exploration of differences in EOL care between the four diagnostic groups

   PELICAN II - Quantitative aims.
3. Assessment of parental perspectives of EOL care in their child/adolescent, including:

   * the development of a new survey instrument (questionnaire)
   * validation and evaluation of psychometric properties of the new survey instrument
4. Exploration of differences in parental perspectives between the four diagnostic groups

   PELICAN II - Qualitative aims.
5. Exploration of parental experiences and needs in their child's EOL care PELICAN II - Mixed methods aims.
6. Explanation and interpretation of quantitative results by exploring parental perspectives of EOL care in their child/adolescent PELICAN III - Quantitative aims.
7. Assessment of formal palliative care education (total hours of training or level A-C according to the European Association of Palliative Care EAPC ), working environment, knowledge and attitudes, and barriers of health care professionals, who are involved in the EOL care of children.

   PELICAN III - Qualitative aims.
8. Exploration of experiences and needs of health care professionals, who are involved in the EOL care of children.

   PELICAN III - Mixed methods aims.
9. Identification and understanding of unmet needs and requirements of health care professionals to provide good quality paediatric EOL care.

ELIGIBILITY:
Inclusion Criteria:

* All children who died in Switzerland in the years 2011 and 2012 due to an oncological, cardiological, neurological condition or during the neonatal phase
* Children and their parents being residents in Switzerland

Exclusion Criteria:

* No mastery of the German, Italian or French language
* Not resident in Switzerland

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between 0-18 years of age dying due to a chronic condition
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Symptom management during the last four weeks of life in dying children aged 0-18 years. | Last 4 weeks of life in dying children
  Outcome measure for PELICAN 1: Description of symptom management of dying children in the last four weeks of life (e.g. pain management, anxiety, delirium).
  Outcome measure for PELICAN 2: Parent's experiences and needs during the End of Life Care of their child (e.g. involvement in decision making processes, consideration of family needs).
  Outcome measure for PELICAN 3:Professional's experiences and needs in Paediatric End of Life Care (e.g. supervision, specialised education).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Cignacco, PD Phd, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Basel, Switzerland

REFERENCES:
- [Background] Eskola K, Bergstraesser E, Zimmermann K, Cignacco E. Paediatric end-of-life care in the home care setting (PELICAN HOME)--a mixed methods study protocol. J Adv Nurs. 2015 Jan;71(1):204-13. doi: 10.1111/jan.12463. Epub 2014 Jun 9. PMID 24909918
- [Background] Zimmermann K, Eskola K, Dorsaz A. [End of life care in pediatrics: when children die]. Krankenpfl Soins Infirm. 2014;107(3):38-9. No abstract available. German. PMID 24683798
- [Background] Bergstraesser E, Zimmermann K, Eskola K, Luck P, Ramelet AS, Cignacco E. Paediatric end-of-life care needs in Switzerland: current practices, and perspectives from parents and professionals. A study protocol. J Adv Nurs. 2015 Aug;71(8):1940-7. doi: 10.1111/jan.12650. Epub 2015 Mar 5. PMID 25740472